CLINICAL TRIAL: NCT02227979
Title: Biological Bases of Individual Variation in Paternal Nurturance
Brief Title: Effects of PURPLE Cry Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, James K. Rilling, PhD, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00044782a
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Shaken Baby Syndrome; Crying; Trauma
MeSH Terms: conditions — Shaken Baby Syndrome; Crying; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): The PURPLE Cry Intervention group will get an 11-page booklet and 12-minute DVD to review.
  Interventions: Behavioral: The Purple Cry Intervention
- Group II (Active Comparator): The control intervention group will get 1 brochure and a DVD on infant safety to review.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: The Purple Cry Intervention — This intervention consists of an 11-page booklet and 12-minute DVD produced by the National Center on Shaken Infant Syndrome.
  Arms: Group I
Behavioral: Control Intervention — This intervention consist of 1 brochure and a DVD on infant safety excerpted from the Safe Start video on infant safety.
  Arms: Group II

SUMMARY:
The proposed study is designed to investigate whether the PURPLE Crying program attains efficacy by optimizing the neural response in the anterior insula, and augmenting activity in regions of the brain known to be important for emotion regulation.

The aim is to determine the effects of the PURPLE Cry Intervention by investigating the following:

* independent variables that may affect a father's neural response to infant cries
* effects of the PURPLE cry intervention, compared to a control intervention, on fathers' reported aversiveness and empathy in response to cry stimuli
* effects of the PURPLE cry intervention, compared to a control intervention, on fathers' neural response to unknown infant cries compared to a tone control
* effects of the PURPLE cry intervention, compared to a control intervention, on fathers' neural responses to own infant cries compared to unknown infant cries

The investigators hypothesize:

* prior to the PURPLE material, fathers' neural responses to infant cry stimuli will be modulated by the following variables: subjective self-reported emotional reaction to cry stimuli, hormone levels, sleep quality and quantity, sex of the infant, infant temperament, life stressors, parental expectations, personality (neuroticism), and father's own childhood experience
* fathers who receive the PURPLE material compared to those that receive the control intervention will report a larger decrease in aversiveness and a larger increase in empathy in response to cry stimuli
* fathers who receive the PURPLE material compared to those that receive the control intervention will show a larger decrease in activity in the anterior insula and amygdala in response to cry stimuli
* fathers who receive the PURPLE material compared to those that receive the control intervention will show a larger increase in activity in regions of the brain important for emotion regulation, such as the dorsolateral prefrontal cortex (PFC) and orbitofrontal PFC
* fathers' neural activity in the amygdala in response to their own infant's cry stimuli will be positively correlated with both their own and infant testosterone levels

DETAILED DESCRIPTION:
40 biological fathers of children age 2 months or younger who are currently cohabitating with the child's mother will be scanned on two separate occasions. The optional second visit will occur after 2 months have passed since the first scan. In the first visit, fathers will receive two MRI scans, one before and one after completing one of the two interventions. Prior to the MRI scan, a blood sample will be collected for measurement of hormone levels. Fathers will be positioned in the MRI scanner where they will receive structural and functional MRI scans of their brain while they listen to auditory stimuli: unknown cries, own cries, and tone controls. Blood sample collection and intervention will not be conducted during the second visit.

ELIGIBILITY:
Inclusion Criteria:

* biological fathers of children age 2 months or younger who are currently cohabitating with the child's mother
* fathers with normal or corrected-to-normal (with contact lenses) vision

Exclusion Criteria:

* history of head trauma, seizures or other neurological disorder
* psychiatric illness
* alcoholism or any other substance abuse
* serious medical illness
* claustrophobia
* ferrous metal in any part of body

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in neural responses to infant cry stimuli | within one visit, pre and post PURPLE intervention, approximately 30 minutes apart
  The effects of the intervention will be assessed by determining changes in neural responses between PURPLE Cry and Brochures treatments from functional magnetic resonance imaging (fMRI)

SECONDARY OUTCOMES:
Change in aversiveness and in empathy | within one visit, pre and post PURPLE intervention, approximately 30 minutes apart
  The effects of the intervention will be assessed by determining changes in aversiveness and in empathy between PURPLE Cry and Brochures treatments by using Davis's Interpersonal Reactivity Index (IRI) and Beck Depression Inventory.
Change in neural activity in the anterior insula and amygdala during unknown infant cry | within one visit, pre and post PURPLE intervention, approximately 30 minutes apart
  The effects of the intervention will be assessed by determining changes in activity in the anterior insula and amygdala between PURPLE Cry and Brochures treatments from functional magnetic resonance imaging (fMRI)
Change in neural activity in the dorsolateral prefrontal cortex (PFC) and orbitofrontal PFC | within one visit, pre and post PURPLE intervention, approximately 30 minutes apart
  The effects of the intervention will be assessed by determining changes in activity in regions of the brain important for emotion regulation between PURPLE Cry and Brochures treatments from functional magnetic resonance imaging (fMRI)
Change in neural activity in the amygdala in response to their own infant's cry stimuli | within one visit, pre and post PURPLE intervention, approximately 30 minutes apart
  The effects of the intervention will be assessed by determining changes in neural activity in the amygdala from functional magnetic resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: James K Rilling, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States